CLINICAL TRIAL: NCT00377702
Title: Epidemiologic Study of Ethnicity and Lifetime Risks for Cardiovascular Disease
Brief Title: Lifetime Risk for Cardiovascular Disease Among Non-White Ethnic Groups
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1350; R21HL085375 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2007-12

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Failure, Congestive; Atrial Fibrillation
Keywords: Coronary Heart Disease; Risk Factors; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Cardiovascular disease (CVD) is one of the leading causes of death in the United States. Currently, there is little information about the lifetime risk of CVD among non-white ethnic groups. This study will analyze data from participants in several ongoing clinical studies to identify the lifetime risk for CVD among various ethnicities.

DETAILED DESCRIPTION:
CVD affects millions of people in the United States. Current treatment guidelines for CVD take into account an individual's risk of developing the disease within 10 years; the intensity of therapy is usually matched to the 10-year risk magnitude. However, many individuals have a low 10-year risk of CVD, but have an elevated lifetime risk of developing the disease. Unfortunately, few studies have examined the lifetime risks for CVD, and these studies have been almost exclusively performed in the Caucasian population. There have been no studies that focus on the lifetime risks for CVD among other ethnic groups. Because the incidence of CVD and other causes of death vary among different ethnic groups, it is important to examine each group separately. Using data from ongoing clinical studies, this study will evaluate the lifetime risks for CVD among different ethnic groups. The results from this study will assist in estimating the future incidence of CVD among ethnic groups, improving risk communication within patient care, and identifying new populations of individuals at risk for CVD.

This study will use previously collected data on 500,000 individuals participating in pre-specified clinical studies. Some of the participating studies include the following: Atherosclerosis Risk in Communities, Framingham Heart, Honolulu Heart, Puerto Rico Heart Health, Coronary Artery Risk Development in Young Adults (CARDIA), Cardiovascular Health, Chicago Heart Association Detection Project in Industry, Women's Health Initiative Observational Studies, and Multiple Risk Factor Intervention Trial (MRFIT). There will be no study visits specifically for this study. Researchers will collect information on CVD risk factors and demographics, including sex, race, and age; they will then compare this information to overall survival, CVD associated survival, and lifetime risk for CVD.

ELIGIBILITY:
Inclusion Criteria:

* Participating in a specified epidemiologic study

Exclusion Criteria:

* Pre-existing CVD prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500000
Dates: Start 2006-07; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald M. Lloyd-Jones, MD, ScM, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Preventive Medicine, Chicago, Illinois, United States